CLINICAL TRIAL: NCT00667901
Title: A Phase 0 Trial of Riluzole in Patients With Resectable Stage III and IV Melanoma
Brief Title: Riluzole in Treating Patients With Stage III or Stage IV Melanoma That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All enrollment, treatment, follow-up & data analysis completed
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James Goydos, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000592958; P30CA072720 (NIH); CINJ-090603; CINJ-IRB-0220060225
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Riluzole; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Immunohistochemistry; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: riluzole
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Riluzole may stop or slow the growth of tumor cells and may be an effective treatment for melanoma.

PURPOSE: This early phase I trial is studying how well riluzole works in treating patients with stage III or stage IV melanoma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the potential effects of glutamate receptor blockade on cellular pathways important in the genesis and progression of melanoma in patients with stage III or IV melanoma undergoing surgical resection.
* To determine whether treatment with riluzole alters expression of activated PLC and ERK in lysates from tumor tissue biopsies.

Secondary

* Determine if treatment with riluzole affects the overall metabolic activity of melanoma tumors as measured by pre- and post-treatment PET scanning, pre- and post-treatment tumor mitotic rate evaluation, and pre- and post-treatment immunohistochemical staining for Ki-67.

OUTLINE: Patients receive oral riluzole twice daily for 14 days. Within 24 hours after the final dose of riluzole, patients undergo standard surgical resection.

Patients undergo tumor tissue sample collection at baseline and during surgery for laboratory studies. Samples are analyzed by routine histology, immunohistochemistry, western blotting, and RT-PCR for Grm1 expression, - RAS and B-raf mutations, PLC and MAP kinase activity, Ki-67 staining, and mitotic rate. Patients also undergo blood sample collection periodically for pharmacokinetics studies.

PET scans are obtained before and after treatment to evaluate the overall metabolic activity of the tumor and how this activity changes with inhibition of the Grm1 pathway.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed melanoma

  * Stage III or IV disease
* Must have at least two resectable tumors or a tumor large enough to undergo pre-treatment core needle biopsy
* Must be eligible for resection of disease with curative or palliative intent

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* ANC ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* AST/ALT ≤ 3 times upper limit of normal (ULN)
* Total bilirubin normal
* Calculated creatinine clearance ≥ 50 mL/min
* INR ≤ 25% of ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 48 hours after completion of study treatment
* No history of allergic reaction to riluzole or similar compounds
* No known history of hepatitis B or C

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the inhibition of components of the Grm1 signaling cascade

SECONDARY OUTCOMES:
Mitoses in nodal metastases and Ki-67 immunostaining (0-3+ scale)

CONTACTS AND LOCATIONS:
Overall Officials: James S. Goydos, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States